CLINICAL TRIAL: NCT04214080
Title: Evaluation of The Effect of Neck and Trunk Stabilization Exercises on Quality of Life and Communication in Children With Cerebral Palsy With Oral Motor Problem
Brief Title: Effect of Trunk Stabilization Exercises on Quality of Life and Communication in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09.2018.337
Record Dates: First submitted 2019-12-16; First posted 2019-12-30 (Actual); Results first posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2018-05

CONDITIONS: Cerebral Palsy
Keywords: Trunk Stabilization Exercises; Oral Motor; Quality of Life; Communication
MeSH Terms: conditions — Cerebral Palsy; Communication

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (SG) (Experimental): In addition to feeding and oral motor intervention strategies, intensive neck and trunk stabilization exercises based on Neurodevelopmental treatment-Bobath (NDT-B) concept principles were applied to this group.
  Treatments were continued 2 days a week for 6 weeks (12 sessions).
  Interventions: Other: Neurodevelopmental treatment (NDT); Other: Feeding and oral-motor intervention strategies; Other: Neck and trunk stabilization exercises
- Control Group (CG). (Placebo Comparator): (NDT-B) concept approaches and feeding and oral motor intervention strategies were applied to this group in routine treatment.
  Treatments were continued 2 days a week for 6 weeks (12 sessions).
  Interventions: Other: Neurodevelopmental treatment (NDT); Other: Feeding and oral-motor intervention strategies

INTERVENTIONS:
Other: Neurodevelopmental treatment (NDT) — NDT is a holistic and interdisciplinary clinical practice model informed by current and evolving research that emphasizes individualized therapeutic handling based on movement analysis for habilitation and rehabilitation of individuals with neurological pathophysiology.
Other: Feeding and oral-motor intervention strategies — Feeding and oral-motor intervention strategies have been developed to address difficulties with sucking, chewing, swallowing, and improve oral-motor skills.
Other: Neck and trunk stabilization exercises — Trunk control affects head control. After gaining head control, it causes jaw stability and oral motor control (tongue control and lip closure). All of these affect communication and quality of life.
  Arms: Study Group (SG)

SUMMARY:
To investigate the effectiveness of neck and trunk stabilization exercises on communication and quality of life (QoL) in children with cerebral palsy (CP) with oral motor problems. Children with CP were randomly divided into Study Group (SG) and Control Group (CG). Neurodevelopmental treatment (NDT) approaches and oral motor therapy were applied to both groups. SG also received neck-trunk stabilization training.

DETAILED DESCRIPTION:
In the multidisciplinary approach, special approaches to secondary problems, oral-motor trainings and communication studies are used in addition to Neurodevelopment treatment approach in the treatment of children with CP. Because of their impact on postural control, neck-trunk stabilization exercises are very important for therapeutic interventions designed to improve quality of life with activities of daily living.

As the increases in neck muscle strength are related to trunk stabilization, trunk stabilization exercises are thought to have positive effects on neck muscle strength. In addition, since the neck and trunk are complementary to each other, it is supported by the literature that neck stabilization exercises and trunk stabilization exercises should be applied together.

ELIGIBILITY:
Inclusion Criteria:

* 1.5 years and older,
* Lack of cooperation problem to prevent communication,
* To have been diagnosed with cerebral palsy and admitted to the hospital for routine control,
* Volunteer to participate in the research,
* Existence of at least one of the items of the "Key Questions" interrogation system showing feeding/swallowing problems in children with cerebral palsy.

Exclusion Criteria:

* Presence of severe vision and hearing loss,
* Use any pharmacological agent to inhibit spasticity,
* He/she had undergone orthopedic surgery or Botulinum Toxin-A injection in the last six months.

Ages: 18 Months to 54 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Ejraei, bachelor, Principal Investigator — Marmara University; Aysel Yıldız Ozer, Assoc. Prof., Study Chair — Marmara University
Locations (1):
- Marmara University Faculty of Health Sciences, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferluga ED, Archer KR, Sathe NA, Krishnaswami S, Klint A, Lindegren ML, McPheeters ML. Interventions for Feeding and Nutrition in Cerebral Palsy [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2013 Mar. Report No.: 13-EHC015-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK132442/ PMID 23596639
- [Background] Shin JW, Song GB, Ko J. The effects of neck and trunk stabilization exercises on cerebral palsy children's static and dynamic trunk balance: case series. J Phys Ther Sci. 2017 Apr;29(4):771-774. doi: 10.1589/jpts.29.771. Epub 2017 Apr 20. PMID 28533628
- [Background] Arvedson JC. Feeding children with cerebral palsy and swallowing difficulties. Eur J Clin Nutr. 2013 Dec;67 Suppl 2:S9-12. doi: 10.1038/ejcn.2013.224. PMID 24301008
- See also: The NDT/Bobath (Neuro-Developmental Treatment/Bobath) Definition. — https://www.ndta.org/
- See also: International Bobath Instructors Training Association — https://ibita.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group (CG).: (NDT-B) concept approaches and feeding and oral-motor intervention strategies were applied to this group in routine treatment.
  Treatments were continued 2 days a week for 6 weeks (12 sessions).
  Neurodevelopmental treatment: NDT is a holistic and interdisciplinary clinical practice model informed by current and evolving research that emphasizes individualized therapeutic handling based on movement analysis for habilitation and rehabilitation of individuals with neurological pathophysiology.
  Feeding and oral-motor intervention strategies: Feeding and oral-motor intervention strategies have been developed to address difficulties with sucking, chewing, swallowing, and improve oral-motor skills.
- Study Group (SG): In addition to feeding and oral-motor intervention strategies, intensive neck and trunk stabilization exercises based on Neurodevelopmental treatment-Bobath (NDT-B) concept principles were applied to this group.
  Treatments were continued 2 days a week for 6 weeks (12 sessions).
  Neurodevelopmental treatment: NDT is a holistic and interdisciplinary clinical practice model informed by current and evolving research that emphasizes individualized therapeutic handling based on movement analysis for habilitation and rehabilitation of individuals with neurological pathophysiology.
  Feeding and oral-motor intervention strategies: Feeding and oral-motor intervention strategies have been developed to address difficulties with sucking, chewing, swallowing, and improve oral-motor skills.
  Neck and trunk stabilization exercises: Trunk control affects head control. After gaining head control, it causes jaw stability and oral motor control (tongue control and lip closure).
Period: Overall Study
Arm/Group | Control Group (CG). | Study Group (SG)
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group (SG) | Control Group (CG). | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Customized [Count of Participants; unit: Participants]
  Age range: (18-48 months) < | 13 | 14 | 27
  Age range: ≥ (48 months) | 7 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 8 | 11 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 20 | 19 | 39
  Syria | 0 | 1 | 1
Cerebral Palsy type [Count of Participants; unit: Participants]
  diplegic | 3 | 1 | 4
  hemiplegic | 2 | 2 | 4
  quadriplegic | 8 | 10 | 18
  hypotonic | 6 | 5 | 11
  dyskinetic | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS)
Description: With VAS, families were asked to mark their communication status with their children. The definitions of the parameter to be evaluated are written on both ends of a 100 mm line. (0= no communication; 10= best communication). According to scale, the higher scores mean a better communication status
Time Frame: Change from VAS was assessed in 0 week (Baseline, in the first session), 6. week (6 weeks after treatment, in the 12th session).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group (SG) | Control Group (CG).
Number analyzed (Participants) | 20 | 20
units on a scale | 6.75 (3.10) | 5.29 (3.33)

2. Primary Outcome: Katz Index of Independence in Activities of Daily Living (ADL)
Description: Measures the capacity of a child to perform the activities that he/she has to do frequently in his/her daily life. The index has 6 questions. The patient gets 1 point if he/she makes each item independently; 0 points if he/she makes dependent. In the total score, 6 points indicate that patient is independent and 0 points indicate that patient is fully dependent. Higher Katz Index score means the better Activities of Daily Living.
Time Frame: Change from Katz was assessed in 0 week (Baseline, in the first session), 6. week (6 weeks after treatment, in the 12th session).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Group (SG) | Control Group (CG).
Number analyzed (Participants) | 20 | 20
score on a scale | 0.70 (1.26) | 0.55 (1.39)

3. Primary Outcome: Pediatric Quality of Life Inventory (PedsQL). Version 4.0- Parent Report for Toddlers (Ages 2-4)
Description: It is a quality of life scale that measures health-related quality of life of children. It consists of 21 items. Items are scored between 0-100. The higher total score means a better health-related quality of life.
Time Frame: Change from PedsQL was assessed in 0 week (Baseline, in the first session), 6. week (6 weeks after treatment, in the 12th session).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Group (SG) | Control Group (CG).
Number analyzed (Participants) | 20 | 20
score on a scale | 48.42 (18.33) | 53.48 (20.28)

4. Primary Outcome: Short Form 36 Questionnaire (SF-36)
Description: Quality of life of mothers was assessed by using the short form 36 questionnaire. It evaluates 8 sub-parameters, consisting of 36 items. 0= poor quality of life; 100= good quality of life. The higher score means a better health-related quality of life
Time Frame: Change from SF-36 was assessed in 0 week (Baseline, in the first session), 6. week (6 weeks after treatment, in the 12th session).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Group (CG).: (NDT-B) concept approaches and feeding and oral motor intervention strategies were applied to this group in routine treatment.
  Treatments were continued 2 days a week for 6 weeks (12 sessions).
  Neurodevelopmental treatment (NDT): NDT is a holistic and interdisciplinary clinical practice model informed by current and evolving research that emphasizes individualized therapeutic handling based on movement analysis for habilitation and rehabilitation of individuals with neurological pathophysiology.
  Feeding and oral-motor intervention strategies: Feeding and oral-motor intervention strategies have been developed to address difficulties with sucking, chewing, swallowing, and improve oral-motor skills.
Arm/Group | Study Group (SG) | Control Group (CG).
Number analyzed (Participants) | 20 | 20
score on a scale | 80.25 (26.97) | 81.75 (17.93)

5. Primary Outcome: Viking Speech Scale (VSS)
Description: This scale has been developed to classify children's speech production. The scale has 4 levels. (Level 1= Speech is not affected by motor disorder; 4= No understandable speech). The low scores mean good speech production.
Time Frame: Change from VSS was assessed in 0 week (Baseline, in the first session), 6. week (6 weeks after treatment, in the 12th session).
Population: We applied this scale in 13 cases (7 in Study group and 6 in Control group). This scale can only be used for patients with SP in age of 4 and above. Therefore, these 13 cases were between the ages of 4-4.5 and provided sufficient age criteria to apply the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Group (SG) | Control Group (CG).
Number analyzed (Participants) | 7 | 6
score on a scale | 3.14 (1.06) | 3.50 (0.837)

6. Primary Outcome: Gross Motor Function Classification System (GMFCS)
Description: The gross motor function of children with cerebral palsy can be categorised into 5 different levels for the clear description of a child's current motor function. The higher level in GMFCS, means a worse and severe outcome. (Level I = Children walk without any limits; Level V= Children are limited in their ability to maintain antigravity head and trunk postures and control leg and arm movements). The low levels means good motor function.
Time Frame: Immediately before the intervention, the evaluation was performed in the first session (only one time).
Measure: Count of Participants; unit: Participants
Groups:
- Study Group (SG): In addition to feeding and oral-motor intervention strategies, intensive neck and trunk stabilization exercises based on Neurodevelopmental treatment-Bobath (NDT-B) concept principles were applied to this group.
  Treatments were continued 2 days a week for 6 weeks (12 sessions).
  Neurodevelopmental treatment: NDT is a holistic and interdisciplinary clinical practice model informed by current and evolving research that emphasizes individualized therapeutic handling based on movement analysis for habilitation and rehabilitation of individuals with neurological pathophysiology.
  Feeding and oral-motor intervention strategies: Feeding and oral-motor intervention strategies have been developed to address difficulties with sucking, chewing, swallowing, and improve oral-motor skills.
  Neck and trunk stabilization exercises: Trunk control affects head control. After gaining head control, it causes jaw stability and oral motor control (tongue control and lip closure). All of these
Arm/Group | Study Group (SG) | Control Group (CG).
Number analyzed (Participants) | 20 | 20
Participants
  level 1 | 4 | 2
  level 2 | 0 | 0
  level 3 | 2 | 0
  level 4 | 4 | 4
  level 5 | 10 | 14

7. Primary Outcome: Communication Function Classification System (CFCS)
Description: CFCS provides 5 levels (CFCS I, II, III, IV, V) to describe everyday communication performance. The higher level in CFCS means a worse and severe outcome. Level 1= effective sender and receiver with unfamiliar and familiar partners; level 5=seldom effective sender and receiver even with familiar partners.
  Low levels mean good communication performance
Time Frame: Immediately before the intervention, an evaluation was performed in the first session (only one time).
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group (SG) | Control Group (CG).
Number analyzed (Participants) | 20 | 20
Participants
  level 1 | 1 | 1
  level 2 | 4 | 3
  level 3 | 8 | 2
  level 4 | 4 | 6
  level 5 | 3 | 8

ADVERSE EVENTS:
Time Frame: 6 weeks.
Arm/Group | Study Group (SG) | Control Group (CG).
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
The limitations of this study are small sample size and relatively short follow-up time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT04214080/Prot_000.pdf
  • Informed Consent Form (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT04214080/ICF_001.pdf
  • Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/80/NCT04214080/SAP_002.pdf